CLINICAL TRIAL: NCT04691388
Title: An Open-Label, Single-Arm, Phase II Trial of Sintilimab Combined With Anlotinib For Metastatic Non-Small Cell Lung Cancer After First-Line PD-1 Inhibitor
Brief Title: A Trial of Sintilimab Plus Anlotinib For Metastatic NSCLC After First-Line PD-1 Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry); Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Yu Xinmin, Chief physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2020-246
Record Dates: First submitted 2020-12-11; First posted 2020-12-31 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: NSCLC
Keywords: sintilimab; anlotinib; NSCLC
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sintilimab +anlotinib (Experimental)
  Interventions: Drug: sintilimab combined with anlotinib

INTERVENTIONS:
Drug: sintilimab combined with anlotinib — All patients will receive sintilimab combined with anlotinib every 3 weeks

SUMMARY:
The combination of immunocheckpoint inhibitors and anti-angiogenesis therapy has synergistic anti-tumor effect and is a reasonable method to improve the prognosis of patients. Therefore, in this study, it is hoped that sintilimab combined with anlotinib can overcome immunotherapy resistance, improve the efficacy of immunotherapy, and further improve the survival of patients, so as to provide more clinical evidence for the treatment of advanced NSCLC patients with negative driver gene after first-line treatment with anti-PD-1 antibody.

DETAILED DESCRIPTION:
Most cancer cells that do not respond to a single immune checkpoint inhibitor escape through the innate immune escape mechanism, allowing them to grow and survive. Different from the inherent resistance mechanism, some patients who initially responded to immune checkpoint inhibitors developed disease progression after a period of treatment and follow-up, suggesting acquired resistance. Therefore, clinical strategies continue to be applied to overcome inherent and acquired resistance to improve the clinical efficacy of immune checkpoint inhibitors. Combining an immune checkpoint inhibitor with another drug that has both immune regulation and anti-tumor properties can enhance the anti-tumor efficacy of any one drug when used alone. Studies have shown that tumor angiogenesis participates in anti-tumor immune regulation and will aggravate the tumor immunosuppressive microenvironment, and anti-angiogenesis therapy can normalize the abnormal vascular structure and function of tumors, and help the recruitment and infiltration of effector T cells. , Reduce the accumulation of immunosuppressive regulatory T cells, relieve the immunosuppressive state, thereby improving the efficacy of immunotherapy. The combination of anti-angiogenic drugs and immune checkpoint inhibitors has become a promising treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participated in this study and signed an informed consent form;
2. Gender is not limited, 18-75 years old; ECOG PS score: 0~1; The expected survival time is more than 3 months;
3. It is diagnosed as advanced (stage IV) non-small cell lung cancer by cytology or histology, and the disease has progressed after receiving PD-1 antibody treatment in the past. According to RECIST 1.1, the efficacy evaluation standard for solid tumors, it has measurable lesions;
4. Provide detectable specimens (tissue or cancerous pleural effusion) for genotype testing before enrollment, and patients whose EGFR, ALK and ROS1 gene test results are all negative;
5. The main organ functions meet the following criteria within 7 days before treatment:

   a) Blood routine examination standard (under no blood transfusion within 14 days):
   * Hemoglobin (HB) ≥9g/dL; ② The absolute value of neutrophils (ANC) ≥ 1.5×109/L;

     ③ Platelet (PLT) ≥80×109/L b) The biochemical inspection shall meet the following standards:
   * Serum total bilirubin (TBIL) ≤ 1.5 × ULN (for patients with Gilbert syndrome, ≤ 3 × ULN); ② Alanine aminotransferase (ALT) and aspartate aminotransferase AST≤2.5ULN, such as liver metastasis, ALT and AST≤5ULN; ③ Serum creatinine (Cr)≤1.5ULN or creatinine clearance rate (CCr)≥50ml/min; c) Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%) d) Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT)≤1.5×ULN;
6. Women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; serum or urine pregnancy tests are negative within 7 days before study entry, And must be a non-lactating patient; men should agree to use contraceptive measures during the study period and within 6 months after the end of the study period;

Exclusion Criteria:

1. Small cell lung cancer (including mixed small cell lung cancer and non-small cell lung cancer);
2. Previously received Anlotinib hydrochloride treatment and other immunotherapy: including but not limited to anti-CTLA-4 antibody, anti-OX40 antibody and anti-CD137 antibody treatment and other immunotherapy;
3. Those who have previously received sunitinib, sorafenib, famitinib, apatinib, regorafenib and other similar VEGFR-TKI small molecule drugs;
4. Imaging (CT or MRI) shows that the tumor focus is ≤ 5 mm from the large blood vessels, or there is a central type tumor that invades the local large blood vessels; or there is obvious lung cavity or necrotic tumor;
5. Untolerable toxicity in previous anti-PD-1/PD-L1 treatments is defined as follows:

1) ≥Level 3 AE related to anti-PD-1/PD-L1; 2) ≥Level 2 immune-related AEs related to anti-PD-1/PD-L1, but AEs that have been relieved or well-controlled after suspension of anti-PD-1/PD-L1 or steroid therapy are not excluded. Past colitis, encephalitis, myocarditis, hepatitis, uveitis and non-infectious pneumonia are excluded; 3) Any level of CNS or eye AE related to anti-PD-1/PD-L1; Note: Patients with previous endocrine AEs can be admitted to the group if they can be stable and asymptomatic under appropriate replacement therapy.

4) Severe hypersensitivity after administration of other monoclonal antibodies; 6. Medical history and comorbidities

1. Patients with active and symptomatic brain metastases, cancerous meningitis, spinal cord compression, or brain or pia mater diseases found in imaging CT or MRI during screening (brain with stable symptoms and treatment completed 28 days before enrollment) Patients with metastases can be included in the group, but they need to be evaluated by MRI, CT or venography to confirm that they have no symptoms of cerebral hemorrhage);
2. Patients with a history of malignant tumors, basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or cervical cancer in situ that have undergone possible curative treatment and have not recurred within 5 years after the start of treatment are excluded;
3. There is any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; subjects need bronchodilators for medical treatment Interventional asthma cannot be included); however, the following patients are allowed to be included in the group: vitiligo, psoriasis, alopecia, well-controlled type I diabetes that do not require systemic treatment, and hypothyroidism with normal thyroid function after replacement therapy;
4. It is necessary to use immunosuppressive agents or systemic therapy to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other curative hormones), and continue to use within 2 weeks of the first administration;
5. Within 4 weeks before the first administration, any patients with bleeding or bleeding event ≥ CTCAE Grade 3, or unhealed wounds, ulcers or fractures;
6. Those who have previously received radiotherapy, chemotherapy, or surgery, after the completion of the treatment (last medication), less than 4 weeks from the first administration, less than 5 drug half-lives of oral targeted drugs; or less than 14 days of oral fluorouracil drugs, mitogen Those who have been less than 6 weeks of C and nitrosourea; those whose adverse events (except for hair loss) caused by previous treatment have not recovered to ≤ CTCAE 1 degree;
7. Abnormal blood coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 ULN), have bleeding tendency or are receiving therapeutic thrombolysis or anticoagulation therapy; Note: in prothrombin The use of anticoagulant drugs for preventive purposes is permitted provided that the international normalized ratio of time (INR) ≤ 1.5.
8. Renal insufficiency: Urine routine test indicates urine protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g;
9. Uncontrollable hypertension (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg, despite the best medical treatment);
10. Unstable angina, myocardial infarction, grade ≥2 congestive heart failure, or arrhythmia requiring treatment (including QTc≥480ms) occurred within 6 months of the first administration;
11. Active or uncontrolled serious infection (≥CTC AE grade 2 infection);
12. Liver cirrhosis, decompensated liver disease, active hepatitis* or chronic hepatitis require antiviral treatment;

    * Active hepatitis (hepatitis B reference: HBsAg positive, and the HBV DNA test value exceeds the upper limit of normal; hepatitis C reference: HCV antibody positive, and the HCV virus titer test value exceeds the upper limit of normal);
13. HIV positive or active tuberculosis;
14. Diabetes is poorly controlled (fasting blood glucose ≥ CTCAE level 2);
15. Have received a preventive vaccine or attenuated vaccine within 4 weeks before the first administration;
16. Subjects who have undergone major surgery or severe trauma have had less than 14 days of elimination of the effects of surgery or trauma before enrollment;
17. Severe cardiovascular disease: Myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmia (including QTc interval ≥450 ms for men and ≥470 ms for women); according to NYHA standards, grade Ⅲ～Ⅳ Insufficiency, or cardiac color Doppler ultrasound examination reveals that the left ventricular ejection fraction (LVEF) is less than 50%;
18. Peripheral neuropathy with ≥CTCAE degree 2 currently exists, except for trauma;
19. Respiratory syndrome (≥CTC AE Grade 2 dyspnea), serous effusion (including pleural fluid, ascites, and pericardial effusion) that need treatment;
20. There are factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
21. Clinically significant hemoptysis (more than 50ml of hemoptysis per day) occurred within 3 months before enrollment; or significant clinically significant bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood at baseline ++ and above, or suffer from vasculitis, etc.;
22. Arterial/venous thrombosis events that occurred within 6 months, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
23. Participated in other anti-tumor drug clinical trials within 4 weeks before enrollment or planned systemic anti-tumor therapy within 4 weeks before grouping or during this study medication period, including cytotoxic therapy, signal transduction inhibitor, immunotherapy ( Or have used mitomycin C) within 6 weeks before receiving the trial drug treatment. Expansion-field radiotherapy (EF-RT) within 4 weeks before grouping or limited-field radiotherapy for tumor lesions to be assessed within 2 weeks before grouping; 7. According to the judgment of the investigator, the patient may have other factors that may cause the study to be terminated halfway, such as other serious diseases or severe laboratory abnormalities or other factors that will affect the safety of the subjects, or test data And the family or society of the sample collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 4 weeks
  ORR assessed by the investigator, including proportions of complete and partial response;

SECONDARY OUTCOMES:
Overall Survival | 5 year
  OS assessed by the investigator
Progression Free Survival | 2 year
  PFS assessed by the investigator
Disease Control Rate | 1 year
  DCR assessed by the investigator
Adverse events | 1 year
  Adverse events (AE), clinical laboratory numerical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Xinmin Yu, doctor, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi X, Lin C, Lou L, He Q, Lou G, Hong W, Shao L, Zhao J, Gu C, Yu X, Jin Y. An Open-Label, Single-Arm, Phase II Trial of Sintilimab Plus Anlotinib for Metastatic Non-Small Cell Lung Cancer After First-Line PD-(L)1 Inhibitor. Cancer Med. 2025 Sep;14(17):e71191. doi: 10.1002/cam4.71191. PMID 40908570